CLINICAL TRIAL: NCT00959699
Title: A Phase 2b, Safety and Efficacy Study of Boceprevir in Patients Coinfected With HIV and Hepatitis C (Protocol No. P05411)
Brief Title: A Phase 2b, Safety and Efficacy Study of Boceprevir in Patients Coinfected With HIV and Hepatitis C (P05411 AM4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05411; MK-3034-025 (Other: Merck study number)
Record Dates: First submitted 2009-07-29; First posted 2009-08-17 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections; Hepatitis C; HCV Infection
Keywords: coinfection; protease inhibitor; HIV
MeSH Terms: conditions — HIV Infections; Hepatitis C; Coinfection | interventions — peginterferon alfa-2b; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PegIFN-2b + RBV (Placebo Comparator): PegIFN-2b (1.5 µg/kg/week subcutaneously) plus RBV (600-1400 mg/day, orally, divided into two daily doses) for 4 weeks followed by placebo to boceprevir plus PegIFN-2b/RBV for 44 weeks with 24 weeks post-treatment follow-up (Control Arm). Participants who do not achieve HCV-RNA <9.3 IU/mL by Treatment Week 24 (TW24) are eligible to cross-over and receive boceprevir along with the PegIFN-2b and RBV for up to 44 weeks.
  Interventions: Drug: PegIFN-2b; Drug: RBV; Drug: Placebo to Boceprevir
- PegIFN-2b + RBV + Boceprevir (Active Comparator): PegIFN-2b (1.5 µg/kg/week subcutaneously) plus RBV (600- 1400 mg/day, orally, divided into two daily doses) for 4 weeks followed by boceprevir (800 mg, orally, 3 times per day) plus PegIFN-2b/RBV for 44 weeks with 24 weeks post-treatment follow-up.
  Interventions: Drug: PegIFN-2b; Drug: RBV; Drug: Boceprevir

INTERVENTIONS:
Drug: PegIFN-2b — PegIFN-2b (1.5 μg/kg/week subcutaneously)
  Other Names: SCH 054031; MK-4031; Pegylated interferon alfa-2b; Peginterferon alfa-2b
Drug: RBV — Ribavirin (600-1400 mg/day, orally, divided into two daily doses)
  Other Names: Ribavirin
Drug: Placebo to Boceprevir — Placebo to boceprevir (orally, three times per day)
  Arms: PegIFN-2b + RBV
Drug: Boceprevir — Boceprevir (800 mg, orally, three times per day)
  Other Names: SCH 503034; MK-3034; Victrelis
  Arms: PegIFN-2b + RBV + Boceprevir

SUMMARY:
The primary objective of this trial is to compare the efficacy of boceprevir (SCH 503034) 800 mg three times a day (TID) orally (PO) in combination with peginterferon alfa-2b (PegIFN-2b) 1.5 µg/kg weekly (QW) subcutaneously (SC) plus weight-based dosing (WBD) of ribavirin (RBV) (600 mg/day to 1400 mg/day) PO to therapy with PegIFN-2b + RBV alone in adult participants coinfected with human immunodeficiency virus (HIV) and previously untreated chronic hepatitis C virus (HCV) genotype 1.

Boceprevir is a potent, orally administered, novel serine protease inhibitor, specifically designed to inhibit the HCV nonstructural protein 3 (NS3) protease and, thereby, inhibit viral replication in HCV-infected host cells. The mechanism of inhibition represents a new mechanism of action compared to both interferon alfa and ribavirin. Based on previous experience with PegIFN-2b and RBV in combination with boceprevir in the HCV-monoinfected population, this combination treatment is expected to provide significant benefit to the HIV/HCV coinfected population. Given the high unmet medical need of these participants and the benefit of the addition of boceprevir to PegIFN-2b/RBV, it is important to demonstrate the safety and efficacy of boceprevir in combination with PegIFN-2b/RBV in participants coinfected with HIV/HCV.

This is a randomized, multi-center trial, double-blinded for boceprevir or placebo in combination with open-label PegIFN-2b/RBV in participants coinfected with HIV and previously untreated chronic HCV (genotype 1), to be conducted in conformance with Good Clinical Practice (GCP). This trial consists of two arms, one control arm (Arm 1) and one experimental arm (Arm 2). Participants in the control arm (Arm 1) may receive boceprevir/PegIFN-2b/RBV via a crossover arm.

ELIGIBILITY:
Inclusion Criteria:

* >=18 and <=65 years of age
* Body weight >=40 and <=125 kg
* Documented history of HIV infection for greater than 6 months prior to Day 1
* On an optimized anti-retroviral treatment regimen (OTR) with stable HIV disease with CD4 >=200 cells/µL and HIV-1 RNA viral load <50 copies/mL
* Documented chronic hepatitis C (CHC) genotype 1 infection (greater than 6 months prior to Day 1)
* Use of acceptable methods of contraception 2 weeks prior to Day 1 and at least 6 months or longer after treatment
* Liver biopsy with histology consistent with CHC and no other etiology

Exclusion Criteria:

* Participants who received prior treatment for hepatitis C other than herbal remedies except those with known hepatotoxicity
* Coinfected with hepatitis B virus (Hepatitis B surface antigen (HBsAg) positive) and/or demonstrating signs and symptoms consistent with concomitant infection
* Evidence of decompensated liver disease
* Participants who have changed their anti-retroviral regimen within the last 3 months prior to Day 1 or had first initiated anti-retroviral therapy within the last 6 months prior to Day 1
* Use of certain HIV medications will not be allowed. Medications will be reviewed by the Investigator
* History of clinically significant opportunistic infections (except oral thrush) within the last year prior to Day 1
* Current evidence of substance abuse within 3 years of the Screening Visit
* History of a clinical diagnosis within the past 6 months of substance abuse prior to Day 1
* Participants receiving opiate agonist substitution therapy but not enrolled in an opiate substitution maintenance program
* History of marijuana use deemed excessive by the Investigator
* Infected with HIV-2
* Use of any HIV protease inhibitor without the coadministration of ritonavir within one month of Day 1 and throughout the period of the trial
* Participants receiving any of the following medication(s) within 2 weeks prior to the Day 1 visit: alfuzosin, antiarrhythmics (amiodarone, bepridil, flecainide, propafenone, and quinidine), ergot derivatives, cisapride, lovastatin, simvastatin, pimozide, triazolam, and orally administered midazolam.

Key Laboratory Exclusion Criteria:

* Hematologic, biochemical, and serologic criteria (growth factors may not be used to achieve trial entry requirements):

  * Hemoglobin <11 g/dL for females and <12 g/dL for males
  * Neutrophils <1500/mm^3 (blacks/African-Americans: <1200/mm^3)
  * Platelets <100,000/mm^3
  * Direct bilirubin >1.5 x ULN (upper limit of normal) of the laboratory reference range. Total bilirubin >1.6 mg/dL unless history of Gilbert's disease or antiretroviral regimen contains atazanavir. If Gilbert's disease is the proposed etiology, this must be documented in the participant's chart
* Alpha fetoprotein (AFP):

  * AFP >100 ng/mL OR
  * AFP 50 to 100 ng/mL (requires a liver ultrasound and participants with findings suspicious for hepatocellular carcinoma are excluded)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Sulkowski M, Pol S, Mallolas J, Fainboim H, Cooper C, Slim J, Rivero A, Mak C, Thompson S, Howe AY, Wenning L, Sklar P, Wahl J, Greaves W; P05411 study investigators. Boceprevir versus placebo with pegylated interferon alfa-2b and ribavirin for treatment of hepatitis C virus genotype 1 in patients with HIV: a randomised, double-blind, controlled phase 2 trial. Lancet Infect Dis. 2013 Jul;13(7):597-605. doi: 10.1016/S1473-3099(13)70149-X. Epub 2013 Jun 12. PMID 23768747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant in the pegylated interferon alfa-2b (PegIFN-2b) + ribavirin (RBV) + boceprevir group withdrew from the study after randomization but prior to administration of any study treatment.
Period: Treatment Period
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Started | 34 | 65
Treated | 34 | 64
Completed | 11 (At TW24, 4 participants not achieving undetectable HCV-RNA crossed-over and received boceprevir.) | 40
Not Completed | 23 | 25
Not completed — Adverse Event | 3 | 13
Not completed — Lack of Efficacy | 15 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Non-Compliance with Protocol | 0 | 1
Not completed — Did not receive treatment | 0 | 1
Not completed — Futility/crossover to boceprevir | 4 | 0
Period: Follow-up Period
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Started | 33 (1 participant didn't enter Follow-up; participants discontinuing treatment could enter Follow-up.) | 62 (2 participants didn't enter Follow-up; participants discontinuing treatment could enter Follow-up.)
Completed | 27 | 56
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir | Total
Number analyzed (Participants) | 34 | 64 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.8) | 42.9 (8.3) | 43.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 22 | 46 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Viral Response (SVR) at Follow-up Week 24 (FW24) Among Randomized Participants Who Received At Least One Dose of Trial Medication
Description: SVR24 is defined as undetectable plasma hepatitis C virus ribonucleic acid (HCV-RNA) at 24 weeks after the end of all study treatment. If there was no value in the FW24 visit window, the closest value available chronologically after this window was used; if a value was still missing after that, the value from Follow-up Week 12 (FW12) was used. HCV-RNA is detected by a nucleic acid amplification test and the lower limit of detection for this assay is 9.3 IU/mL.
Time Frame: Up to Week 72
Population: All randomized participants receiving at least one dose of any study medication (Full Analysis Set); this includes 3 participants who did not enter the Follow-Up Period.
Measure: Number; unit: percentage of participants
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Number analyzed (Participants) | 34 | 64
percentage of participants | 29.4 [14.1 to 53.3] | 62.5
Statistical Analysis 1: Comparison: PegIFN-2b + RBV vs PegIFN-2b + RBV + Boceprevir; The methodology for 95% Confidence Interval (CI) is based on a Modified Koch approach which adjusted for Randomization Strata of Cirrhosis/Fibrosis (Yes or No). The adjustment of randomization strata of HCV-RNA (< or >= 800,000 IU/mL) was not possible due to sparse data; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel p-value is adjusted for randomization strata of HCV-RNA (< or >= 800,000 IU/mL) and Cirrhosis/Fibrosis (Yes or No); Strata-Adjusted Difference = 33.7, 95% CI 2-sided [14.1 to 53.3]

2. Secondary Outcome: Percentage of Participants Achieving SVR24 Among Randomized Participants Who Received At Least One Dose of Boceprevir (Experimental) or Placebo (Control)
Description: SVR24 is defined as undetectable plasma HCV-RNA 24 weeks after the end of all study treatment. If there was no value in the FW24 visit window, the closest value available chronologically after this window was used; if a value was still missing after that, the value from FW12 was used. HCV-RNA is detected by a nucleic acid amplification test and the lower limit of detection for this assay is 9.3 IU/mL.
Time Frame: Up to Week 72
Population: All randomized participants receiving one dose of boceprevir (PegIFN-2b + RBV + Boceprevir group) or placebo to boceprevir (PegIFN-2b + RBV group), defined as the Modified Intent-to-Treat Population; this includes 2 participants who did not enter the Follow-up Period.
Measure: Number; unit: percentage of participants
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Number analyzed (Participants) | 33 | 62
percentage of participants | 30.3 | 64.5
Statistical Analysis 1: Comparison: PegIFN-2b + RBV vs PegIFN-2b + RBV + Boceprevir; The methodology for 95% CI is based on the asymptotic normal approximation to the binomial distribution; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Observed Difference = 34.2, 95% CI 2-sided [14.5 to 53.9]

3. Secondary Outcome: Percentage of Participants With Early Virologic Response (EVR) Who Achieved SVR24
Description: EVR was defined as undetectable HCV-RNA at Treatment Week (TW) 2, 4, 8, or 12. HCV-RNA was detected by a nucleic acid amplification test and the lower limit of detection for this assay is 9.3 IU/mL.
Time Frame: Up to Week 12
Population: All randomized participants receiving at least one dose of any study medication (Full Analysis Set); this includes 3 participants who did not enter the Follow-Up Period. No participants had undetectable HCV-RNA at Week 2; the "n" value in the table below represents the number of participants with EVR at that time point.
Measure: Number; unit: percentage of participants
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Number analyzed (Participants) | 34 | 64
percentage of participants
  HCV-RNA undetectable at Week 2 (n=0, 0) | 0 | 0
  HCV-RNA undetectable at Week 4 (n=3, 3) | 100 | 100
  HCV-RNA undetectable at Week 8 (n=5, 27) | 100 | 92.6
  HCV-RNA undetectable at Week 12 (n=8, 38) | 87.5 | 92.1

4. Secondary Outcome: Percentage of Participants With Undetectable HCV-RNA at Follow-up Week 12 (FW12)
Description: The virologic response at FW12 was considered SVR12 with an additional rule for handling missing data: participants with missing HCV-RNA assessment at FW12 but having non-missing, undetectable HCV-RNA assessments at both FW4 and FW24, were assumed to be responders for SVR12. HCV-RNA was detected by a nucleic acid amplification test and the lower limit of detection for this assay is 9.3 IU/mL.
Time Frame: Up to Week 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Number analyzed (Participants) | 34 | 64
percentage of participants | 26.5 | 62.5

5. Secondary Outcome: Change From Baseline in log10 HCV-RNA at Treatment Week 4 (TW4)
Description: This is a measure of the change in the amount of HCV-RNA in the plasma at the end of 4 weeks of treatment. HCV-RNA was detected by a nucleic acid amplification test and the lower limit of detection for this assay is 9.3 IU/mL.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Number analyzed (Participants) | 34 | 64
participants
  Participants with <1 positive log drop | 15 | 28
  Participants with >= 1 positive log drop | 16 | 32
  Participants with undetectable HCV-RNA | 3 | 3
  Participants with missing data | 0 | 1

6. Secondary Outcome: Percentage of Participants With HCV Virologic Breakthrough or Incomplete Virologic Response/Rebound
Description: Virologic breakthrough is defined as achieving undetectable HCV-RNA and subsequently having an HCV-RNA level of >1000 IU/mL. Incomplete Virologic Response/Rebound is defined as having a one log10 increase in HCV-RNA from the participant's nadir, with an HCV-RNA >1000 IU/mL. HCV-RNA was detected by a nucleic acid amplification test and the lower limit of detection for this assay is 9.3 IU/mL.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PegIFN-2b + RBV | PegIFN-2b + RBV + Boceprevir
Number analyzed (Participants) | 34 | 64
percentage of participants
  Virologic breakthrough | 0 | 6.3
  Incomplete response | 17.6 | 9.4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through Week 72.
Description: One participant randomized to the boceprevir arm never received study drug.
  Adverse events for the 4 participants who crossed-over to boceprevir treatment at Treatment Week 24 (TW24) are included in the assigned treatment arm (PegIFN-2b + RBV ) until TW24 and are presented separately for the period following the crossover.
Groups:
- PegIFN-2b+RBV: PegIFN-2b (1.5 µg/kg/week subcutaneously) plus RBV (600-1400 mg/day, orally, divided into two daily doses) for 4 weeks followed by placebo to boceprevir plus PegIFN-2b/RBV for 44 weeks with 24 weeks post-treatment follow-up (Control Arm). Participants who do not achieve HCV-RNA <9.3 IU/mL by Treatment Week 24 (TW24) are eligible to cross-over and receive boceprevir along with the PegIFN-2b and RBV for up to 44 weeks.
- PegIFN-2b+RBV+Boceprevir: PegIFN-2b (1.5 µg/kg/week subcutaneously) plus RBV (600- 1400 mg/day, orally, divided into two daily doses) for 4 weeks followed by boceprevir (800 mg, orally, 3 times per day) plus PegIFN-2b/RBV for 44 weeks with 24 weeks post-treatment follow-up.
- Boceprevir Crossover: (After Treatment Week 24) PegIFN-2b (1.5 µg/kg/week subcutaneously) plus RBV (600- 1400 mg/day, orally, divided into two daily doses) plus boceprevir (800 mg, orally, 3 times per day) for up to 44 weeks with 24 weeks post-treatment follow-up.
Arm/Group | PegIFN-2b+RBV | PegIFN-2b+RBV+Boceprevir | Boceprevir Crossover
Serious Adverse Events (participants affected / at risk) | 7/34 | 11/64 | 0/4
Other Adverse Events (participants affected / at risk) | 33/34 | 62/64 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIFN-2b+RBV (N=34) | PegIFN-2b+RBV+Boceprevir (N=64) | Boceprevir Crossover (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VULVAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIFN-2b+RBV (N=34) | PegIFN-2b+RBV+Boceprevir (N=64) | Boceprevir Crossover (N=4)
ANAEMIA (Blood and lymphatic system disorders) | 8 (8) | 26 (40) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 12 (14) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 1 (1)
PALPITATIONS (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
PORPHYRIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 2 (2) | 2 (3) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 6 (7) | 0 (0)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 2 (2) | 5 (6) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 6 (8) | 21 (30) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 11 (12) | 26 (37) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
TONGUE DISCOLOURATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 5 (9) | 18 (23) | 0 (0)
ASTHENIA (General disorders) | 9 (9) | 22 (30) | 2 (2)
CHILLS (General disorders) | 5 (5) | 5 (5) | 0 (0)
FATIGUE (General disorders) | 12 (15) | 25 (35) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 13 (29) | 16 (24) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 1 (1) | 4 (4) | 0 (0)
IRRITABILITY (General disorders) | 5 (5) | 10 (11) | 1 (1)
MALAISE (General disorders) | 2 (2) | 3 (3) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 3 (3) | 0 (0)
PAIN (General disorders) | 1 (1) | 5 (5) | 0 (0)
PYREXIA (General disorders) | 7 (13) | 24 (60) | 1 (1)
FOLLICULITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
GINGIVAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 4 (5) | 6 (7) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 5 (5) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 2 (2) | 3 (5) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 5 (6) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 8 (9) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (6) | 22 (22) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (12) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 8 (9) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 5 (5) | 18 (18) | 2 (2)
HEADACHE (Nervous system disorders) | 6 (6) | 18 (63) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
AFFECT LABILITY (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
ANXIETY (Psychiatric disorders) | 5 (8) | 10 (11) | 0 (0)
APATHY (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 4 (4) | 11 (11) | 0 (0)
DRUG ABUSE (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 9 (12) | 15 (17) | 0 (0)
NERVOUSNESS (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 1 (1) | 5 (5) | 0 (0)
METRORRHAGIA (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (10) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6) | 12 (12) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (11) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (4) | 13 (16) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc.) that report any results of the trial. The sponsor shall have the right to review and comment.